CLINICAL TRIAL: NCT05208021
Title: The Effect of Individual Psychoeducation Program Based on the Health Promotion Model on the Healthy Living Behaviors of Individuals With Schizophrenia
Brief Title: The Effect of Psychoeducation Program on Healthy Living Behaviors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Mahinur Betül Çalışkan, PhD student in nursing departman, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SY200217B08
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia
Keywords: healthy lifestyle; schizophrenia; motivational interviewing; psychiatric nursing
MeSH Terms: conditions — Schizophrenia | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Who Masked: Participant
Masking Description: Experimental: Intervention group "Health Promotion Model and the Motivational Interview-Based Health Protection and Promotion Program was applied to the intervention group No Intervention: Control Group Only data collection was carried out. No attempt was made by the researcher during the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): "Health Promotion Model and the Motivational Interview-Based Health Protection and Promotion Program was applied to the intervention group
  Interventions: Behavioral: Intervention group (Motivational Interviewing)
- Control Group (No Intervention): Only data collection was carried out. No attempt was made by the researcher during the study

INTERVENTIONS:
Behavioral: Intervention group (Motivational Interviewing) — The Health Promotion Model and the Motivational Interview-Based Health Protection and Promotion Program were applied to the experimental group, which consisted of 6 sessions and lasted an average of 60-120 minutes. Sessions were held in the form of individual interviews due to the pandemic and social distance conditions.
  Arms: Intervention group

SUMMARY:
1.031 / 5.000 Çeviri sonuçları This research was planned to determine the effect of health protection and promotion program based on motivational interviewing based on Pender's Health Promotion Model on healthy lifestyle behaviors of individuals with schizophrenia. When the national and international literature is examined, it is known that there are descriptive studies on the physical health of individuals with mental disorders, and interventional intervention programs under the leadership of psychiatric nurses for the protection and development of the physical health of individuals with mental disorders are very limited. In this context, psychiatric nurses act as a bridge between mental and physical health for patients. It is thought that this study, which will be conducted to evaluate the healthy lifestyle behaviors of individuals with schizophrenia, of the Health Promotion Model and motivational interview-based health protection and promotion program will contribute to the literature, provide data for future studies, and be an applicable model for TRSMs.

DETAILED DESCRIPTION:
Research Istanbul Bakirkoy Prof. Dr. In Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital Bakırköy Community Mental Health Center, the experimental research design was carried out with a pretest and posttest control group. The study population of this study consisted of patients aged 18-65 years who were diagnosed with schizophrenia and other psychotic disorders (N=502). The sample of the study consisted of patients diagnosed with schizophrenia and other psychotic disorders who met the sampling criteria determined in the study (n=52). In the Power analysis of the research, the sample size was determined as 2 groups, with 26 people as the experimental group and 26 people as the control group, with a total of 52 people in the 95% confidence interval. In the study, 52 patients diagnosed with schizophrenia and other psychotic disorders who met the sample selection criteria and volunteered to participate in the study were divided into experimental and control groups using simple random sampling technique. As data collection tools in the research; Personal Information Form, Healthy Life Style Behavior Scale II, Health Improvement Profile, Anthropometric Measurements and Vital Findings and Stage of Change Diagnosis Form were used. The implementation of the research was completed in four stages. In the first stage, the "Health Promotion Model and Motivational Interview-Based Health Protection and Promotion Program" was developed by the researcher in line with the literature review. In the second stage, after the program was introduced to all participants who met the inclusion criteria and their written consent was obtained, pre-tests including the variables of the research were applied, and then the participants were assigned to the experimental and control groups by randomization method. Sessions were held in the form of individual interviews due to the pandemic and social distance conditions. In the third stage, the Health Promotion Model and the Motivational Interview-Based Health Protection and Promotion Program were applied to the experimental group, which consisted of 6 sessions and lasted an average of 60-120 minutes to discuss the warm-up period and the main themes of the sessions in each individual session. A summary of the previous session was made to remember what was done in the first 5-10 minutes of each session. "Weekly Nutrition Follow-up Form", "Weekly Step Count Follow-up Form", "Weekly Stress Follow-up Form", "Weekly Leisure Activities Follow-Up Form" and "Weekly Sleep Diary" prepared by the researcher for the experimental group participants were handed over to the patients as homework. They were asked to fill it out weekly and bring it to their next session. No intervention was made to the patients in the control group during the six-week period. During this process, both experimental and control group patients continued their routine treatments including drug treatments, doctor's controls, psychoeducation, individual therapy, and other programs at the Community Mental Health Center. At the end of the sixth session, the measurement tools were applied again and the implementation phase of the research was ended. After the Health Promotion Model and Motivational Interview-Based Health Protection and Improvement Program sessions applied to the experimental group were completed, the post-test was applied three and six months later, and the control group was followed-up by applying the post-test six weeks, three and six months later.

ELIGIBILITY:
Inclusion Criteria:

* Who agrees to participate in the research himself or his guardian,
* Diagnosed with schizophrenia and other psychotic disorders for at least six months according to DSM-V diagnostic criteria,
* Registered with the Community Mental Health Center and coming regularly,
* Between the ages of 18-65,
* Who can read and write Turkish,
* Using antipsychotic medication for at least six months,
* Not in the "pre-thinking" stage in the change cycle stage,
* No skeletal, muscular, nervous system disease that prevents physical activity or healthy eating,
* They are patients without mental retardation, neurocognitive disorder, alcohol or substance abuse.

Exclusion Criteria:

* Failure of himself or his guardian to participate in the research,
* Without a diagnosis of schizophrenia and other psychotic disorders,
* Not coming regularly to the Community Mental Health Center,
* Under 18 years old and over 65 years old,
* Does not speak Turkish,
* Not using regular antipsychotic medication,
* In the "pre-thinking" stage of the cycle of change,
* Those with skeletal, muscular, nervous system diseases that prevent physical activity or healthy nutrition,
* They are patients with mental retardation, neurocognitive disorder, alcohol and substance addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Healthy Life Style Behavior Scale II | 8 month
  Scale; It consists of six sub-factors consisting of spiritual development, interpersonal relations, nutrition, physical activity, health responsibility and stress management and a total of 52 items. The scale is a four-point Likert scale, scored as never: 1, sometimes: 2, often: 3, and regularly: 4.

SECONDARY OUTCOMES:
Health Improvement Profile | 8 month
  The Health Promotion Profile was developed to diagnose the physical health conditions of individuals diagnosed with mental disorders. This profile, which enables physical health risk assessment, is different for men and women. The Health Promotion Profile consists of four sub-dimensions: measurements, blood tests, screenings and lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Mahinur Betül ÇALIŞKAN, MSc, Principal Investigator — Istanbul Saglik Bilimleri University
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No